CLINICAL TRIAL: NCT00453817
Title: Suivi Par résonance magnétique après Transplantation d'îlots de Langerhans
Brief Title: Islet of Langerhans Graft Monitoring by Magnetic Resonance Imaging
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Feasibility issues
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Thierry Berney, Professor of Surgery, University Hospital, Geneva
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 04-019
Record Dates: First submitted 2006-10-04; First posted 2007-03-29 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-12

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: islet transplantation; imaging; graft monitoring; magnetic resonance imaging
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — ferumoxides; Islets of Langerhans Transplantation; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Study subjects (Experimental): One-arm observational study
  Interventions: Drug: ferucarbotran (iron-based MRI contrast agent); Procedure: Islet transplantation; Procedure: Magnetic resonance imaging

INTERVENTIONS:
Drug: ferucarbotran (iron-based MRI contrast agent) — islets will be incubated with ferucarbotran prior to transplantation, for imaging after transplantation
Procedure: Islet transplantation — intraportal percutaneous islet transplantation
Procedure: Magnetic resonance imaging — Magnetic resonance imaging of the liver before and after islet transplantation (6 days, 6 weeks, 6 months, 1 year)

SUMMARY:
The primary objective of this pilot study is to assess the feasibility and safety of ex vivo islet labelling prior to intraportal transplantation in patients with type 1 diabetes with the purpose of islet graft imaging. The secondary objective is to determine the usefulness of this method for long-term islet graft monitoring.

DETAILED DESCRIPTION:
The objectives will be addressed in a pilot study. We plan to enroll 15 patients over 3 years in islet transplantation alone (ITA), islet-after-kidney transplantation (IAK) or simultaneous islet-kidney transplantation (SIK) procedures. Patients will be followed-up for 1 year after transplantation.

Islet isolation and transplantation Islets will be isolated and purified from pancreata harvested from multiorgan donors, according to the automated method described by Ricordi, with local modifications. After isolation, islets will be cultured overnight at 37°C in CMRL medium. After overnight culture, islets will be changed to fresh medium containing carbodextran-coated iron oxide nanoparticles (Resovist; Schering, Baar, Switzerland), at a target concentration of 5ul/ml, with a total dose not exceeding 0.08 ml/kg body weight, and further cultured for a total of 48-72 hours at 25°C until transplantation. Islet transplantation will be performed by intraportal infusion of the islet preparation, using a transhepatic percutaneous approach. Patients will receive infusions of at least 5,000 IEQ/kg. A second islet infusion will be administered to patients who have not reached insulin independence after the first transplant.

Graft monitoring and follow-up Patients will be followed for 1 year after last islet infusion. MRI will be performed prior to, 6 days, 6 weeks, 6 months and 1 year after islet infusion. A standard MRI protocol will be adapted. Since transplanted islets are already iron-labeled, no injection of contrast media will be done during MRI examination, and MRI sequences will not be repeated. After a scout image, axial views of the liver will be acquired with a fast gradient echo T2* weighted sequence, a fast spin echo T2* weighted sequence, ultrashort echo time T2* weighted sequences, a spin echo T1 weighted sequence and in/out of phase fast gradient echo T1 weighted sequences. Iron-labeled islets will be visualized as a loss of signal on fast gradient echo T2* weighted sequence, and the islet mass will be assessed in a semi-quantitative fashion using a visual scale. Finally, ultrashort echo time sequences will be used to generate a T2 map. The amount of iron contained inside the transplanted islets will be quantified based on the T2 map and the correction for the distribution of the iron particles inside the liver.

Monitoring results will be compared to islet function assessed by routine tests: exogenous insulin requirement, C-peptide, HbA1c, fructosamine, arginine stimulation test. Results will be analyzed retrospectively for the first 2 years. According to results of the analysis, the investigators may decide to intervene proactively (i.e. administer antirejection therapy) in the last year of the study, whenever results suggestive of a dysfunction are observed.

ELIGIBILITY:
Inclusion Criteria:

* All patients on the waiting list for an islet of Langerhans transplantation procedure

Exclusion Criteria:

* Allergy to ferucarbotran
* Inability to undergo MRI (patients carrying osteosynthesis material, pacemakers or other metallic devices)
* Claustrophobia (tolerance to MRI)
* Hemosiderosis/hemochromatosis (interference with MRI signal)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2005-06; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Semi-quantitative assessment of intrahepatic MRI signal on T2*-weighted sequences, at 6 days, 6 weeks, 6 months and 1 year after transplantation | 2005-2009

SECONDARY OUTCOMES:
Islet graft function assessed by exogenous insulin requirements, HbA1c, mean amplitude of glucose excursions (MAGE) and fasting C-peptide. | 2005-2009

CONTACTS AND LOCATIONS:
Overall Officials: Thierry Berney, MD, MSc, Principal Investigator — University Hospital, Geneva
Locations (1):
- Geneva University Hospitals Department of Surgery, Geneva, Switzerland